CLINICAL TRIAL: NCT00091598
Title: ARIES 1 and ARIES 2: Ambrisentan in PAH - A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter, Efficacy Study of Ambrisentan in Subjects With Pulmonary Arterial Hypertension
Brief Title: ARIES - Ambrisentan in Patients With Moderate to Severe Pulmonary Arterial Hypertension (PAH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARIES
Expanded Access: Available
Record Dates: First submitted 2004-09-10; First posted 2004-09-14 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2010-03

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — ambrisentan

INTERVENTIONS:
Drug: Ambrisentan

SUMMARY:
The primary objective is to determine the effect of ambrisentan on exercise capacity in subjects with PAH.

DETAILED DESCRIPTION:
ARIES-1 in North America and Australia

ARIES-2 in Western and Eastern Europe, South America and Israel

Subjects in these randomized studies will receive one of two doses of ambrisentan or placebo. Inclusion is not based on a specified WHO functional classification. Rather, subjects with WHO Class I-IV symptoms are eligible if their 6-minute walk distance is 150-450 meters and they meet the study-specified hemodynamic criteria. Subjects with anorexigen or HIV infection related PAH are eligible but subjects with congenital heart disease and pediatric subjects are excluded. The study requires a historical cardiac catheterization and other diagnostic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PAH (formally known as PPH), or PAH associated with collagen vascular disease, anorexigen use, or HIV infection;
* Historical cardiac catheterization with the following hemodynamic criteria:

Mean pulmonary artery pressure greater than or equal to 25 mmHg; Pulmonary vascular resistance greater than 3 mmHg/L/min; Pulmonary capillary wedge pressure or left ventricular end diastolic pressure less than 15 mmHg;

* 6-minute walk distance of at least 150 meters, but no more than 450 meters;
* Total lung capacity greater than or equal to 70% and FEV1 greater than or equal to 65% of predicted normal;

Exclusion Criteria:

* Portopulmonary hypertension;
* Subjects with PAH due to or associated with coronary artery disease, left heart disease, interstitial lung disease, chronic obstructive pulmonary disease, veno-occlusive disease, chronic thromboembolic disease, or sleep apnea;
* Bosentan (Tracleer®), sildenafil (Viagra®), or chronic prostanoid therapy within 4 weeks of screening;
* Serum ALT or AST lab value that is greater than 1.5 times the upper limit of normal;
* Contraindication to treatment with an endothelin receptor antagonist;
* Subject with cardiovascular, hepatic, renal, hematologic, gastrointestinal, immunologic, endocrine, metabolic, or central nervous system disease that may adversely affect the safety of the subject;
* Participation in a clinical study involving another investigational drug within 4 weeks of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372
Dates: Start 2004-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline at Week 12 of six minute walk distance

SECONDARY OUTCOMES:
Change from baseline at Week 12 of:
Borg Dsypnea Index
WHO Functional Classification
SF-36
Time to Clinical Worsening

CONTACTS AND LOCATIONS:
Overall Officials: Lewis J. Rubin, MD, Study Chair — University of California San Diego, San Diego School of Medicine
Locations (46):
- United States (44):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - Brentwood Biomedical Research Institute, Los Angeles, California
  - University of California-Davis, Sacramento, California
  - University of California San Diego Medical Center, San Diego, California
  - Los Angeles County Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Myogen, Westminster, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Mt. Sinai Medical Center, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Loyola University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Ochsner Clinic, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Northshore University/Long Island Jewish Hospital, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - Mt. Sinai Medical Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Cardiology PC, Syracuse, New York
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - St. Paul Hospital, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas - San Antonio, San Antonio, Texas
  - Scott & White Hospital, Temple, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Heart Care Associates, Milwaukee, Wisconsin
- St. Vincent's Hospital, Sydney, New South Wales, Australia
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Galie N, Olschewski H, Oudiz RJ, Torres F, Frost A, Ghofrani HA, Badesch DB, McGoon MD, McLaughlin VV, Roecker EB, Gerber MJ, Dufton C, Wiens BL, Rubin LJ; Ambrisentan in Pulmonary Arterial Hypertension, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Efficacy Studies (ARIES) Group. Ambrisentan for the treatment of pulmonary arterial hypertension: results of the ambrisentan in pulmonary arterial hypertension, randomized, double-blind, placebo-controlled, multicenter, efficacy (ARIES) study 1 and 2. Circulation. 2008 Jun 10;117(23):3010-9. doi: 10.1161/CIRCULATIONAHA.107.742510. Epub 2008 May 27. PMID 18506008
- See also: Pulmonary Hypertension Association — http://www.phassociation.org